CLINICAL TRIAL: NCT01241279
Title: A Two Arm Prospective, Randomized, Double-Masked Clinical Evaluation of Accommodation Measurements After Bilateral Implantation of an Aspheric Accommodating Lens and Monofocal Aspheric Lenses
Brief Title: Accommodation Measurements After Bilateral Implantation of an Aspheric Accommodating Lens and Monofocal Aspheric Lenses
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated due to low enrollment
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 657
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Cataract
Keywords: cataract surgery; intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crystalens AO (Experimental): A silicone multi-piece accommodating intraocular lens
  Interventions: Device: Crystalens AO
- SoftPort LI61AO (Active Comparator): A silicone multi-piece foldable aspheric intraocular lens
  Interventions: Device: SoftPort LI61AO

INTERVENTIONS:
Device: Crystalens AO — Participants will undergo small incision cataract surgery (phacoemulsification). At the time of surgery, eligible participants will be implanted bilaterally with the Crystalens AO intraocular lens.
  Arms: Crystalens AO
Device: SoftPort LI61AO — Participants will undergo small incision cataract surgery (phacoemulsification). At the time of surgery, eligible participants will be implanted bilaterally with the SoftPort LI61AO intraocular lens.
  Arms: SoftPort LI61AO

SUMMARY:
The objective of this study is to demonstrate the correlation of near vision and changes in higher order aberrations following lens extraction and to characterize the defocus curves of Crystalens® AO™ intraocular lens (IOL) versus the monofocal aspheric SofPort® LI61AO IOL in adults.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have clear intraocular media other than cataract.
* Subjects must have a clinically documented diagnosis of age-related bilateral cataracts that are considered amenable to treatment with standard phacoemulsification cataract extraction.
* Subjects must be undergoing primary IOL implantation for the correction of aphakia following central continuous curvilinear anterior capsulorrhexis and phacoemulsification cataract extraction.
* Subjects must require a spherical lens power from 10.00 D to 30.00 D.
* Subjects must be willing and able to return for all scheduled follow-up examinations for each eye from days 1 through 180 following surgery.
* Subjects must have ≤ 1.25 D of preoperative corneal astigmatism.

Exclusion Criteria:

* Subjects with corneal pathology potentially affecting topography.
* Subjects whose fundus cannot be assessed preoperatively.
* Subjects with diagnoses of degenerative visual disorders (eg, macular degeneration, or other retinal disorders) that cause potential acuity losses to a level worse than 20/30 as verified by OCT.
* Subjects with conditions with increased risk of zonular rupture, such as pseudoexfoliation syndrome.
* Subjects who have any active inflammation or edema (swelling) of the cornea, including but not limited to the following: keratitis, keratoconjunctivitis, and keratouveitis.
* Subjects with uncontrolled glaucoma.
* Subjects with previous retinal detachment.
* Subjects with visually significant diabetic retinopathy (proliferative or non-proliferative) which reduces potential acuity to 20/30 or worse.
* Subjects with rubella, bilateral congenital, traumatic, complicated or polar cataract.
* Subjects with marked microphthalmos or aniridia.
* Subjects who have had previous corneal surgery.
* Subjects with irregular corneal astigmatism.
* Subjects with amblyopia which reduces potential acuity to worse than 20/30.
* Subjects with optic atrophy.
* Subjects with iris neovascularization.
* Subjects with clinically significant retinal pigment epithelium/macular changes which reduces potential acuity to 20/30 or worse.
* Subjects with chronic use of systemic steroids or immunosuppressive medications.
* Subjects lacking intact binocular vision.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Varughese, Study Director — Valeant Pharmaceuticals/Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6 subjects (11 eyes) were enrolled at one investigational site in the US. First participant enrolled 10/26/2010; last participant visit 12/01/2011.
Pre-assignment Details: Due to the small sample size, NO STATISTICAL OR CLINICALLY MEANINGFUL CONCLUSIONS RELATED TO THE STUDY ENDPOINTS CAN BE MADE.
Period: Overall Study
Arm/Group | Crystalens AO | SoftPort LI61AO
Started | 4 | 2
Completed | 4 | 1
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crystalens AO | SoftPort LI61AO | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Customized [Number; unit: participants]
  Age 54 to 70 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Amplitude of Accommodation
Description: The measurement of optical change in the power of the eye when viewing from far to near. Accommodation decreases as age increases resulting in an inability to focus on near objects.
Time Frame: Visit 4 (postoperative day 120-180)
Population: DUE TO THE SMALL SAMPLE SIZE, NO STATISTICAL OR CLINICALLY MEANINGFUL CONCLUSIONS RELATED TO THE STUDY ENDPOINTS CAN BE MADE.
Arm/Group | Crystalens AO | SoftPort LI61AO
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Visual Acuity
Description: Number of correct letters on an early treatment diabetic retinopathy study (ETDRS) chart to measure distance visual acuity and the smallest readable print size on an Minnesota Low-Vision Reading (MNREAD) acuity chart for intermediate and near visual acuity (VA). Visual acuity measured in LogMAR.
Time Frame: All visits through visit 4 (day 160-180)
Population: as for outcome 1
Arm/Group | Crystalens AO | SoftPort LI61AO
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | Crystalens AO | SoftPort LI61AO
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2

LIMITATIONS AND CAVEATS:
Study terminated early due to lack of enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee and the Investigator(s) are completed. The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.